CLINICAL TRIAL: NCT07134881
Title: Navigating Advanced Illness Goals And Treatment With Digital Engagement (NAVIGATE): A Randomised Control Trial
Brief Title: Navigating Advanced Illness Goals And Treatment With Digital Engagement (NAVIGATE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Gerald Koh, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ECOS 2025-0194
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Paliative Care; Advance Care Planning; Digital Education Interventions; Values, Social; Goals of Care
Keywords: randomised control trial; digital intervention; advance care planning; goals of care; palliative care

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, participant-level randomised trial. Upon providing consent and completion of the baseline survey, enrolled caregiver participants will be randomly assigned 1:1 to the experimental and comparator arms using the built-in randomizer function in the online survey software (Qualtrics). Balance between the allocation arms will be achieved by stratifying based on illness.
Who Masked: Participant
Masking Description: Treatment allocation will be masked from participants for the entirety of the study. We do not anticipate unblinding of participants to treatment status. Effort to maintain blinding of participants include training our research coordinators (RCs) to strictly follow a protocol and script in all interactions with participants. RCs are blinded of treatment allocation during recruitment, consent-taking and baseline survey process, minimising the risk of selection bias. Once participants are randomised into their allocated arm, RCs will be aware of the participant's treatment allocation as RCs will need to ensure that participants successfully complete the signup process required for the intervention arm. Risks of unmasking caregivers participants is minimal as followup questionnaires are completed via self-administered online survey without the RCs being present.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator arm (Active Comparator): For caregiver participants: Usual care. For patient participants: usual care, as prescribed by the clinical care team, is unaffected by the study design and we only conduct observational measurements of patient participants during the course of the study.
  Interventions: Other: Usual Care
- Intervention arm (Experimental): For caregiver participants: Enrolled caregiver participants randomised in the intervention arm will be directed to the intervention digital website and guided through the signup process. Once logged in, they are asked to explore and use the website contents and tools in their own time.
  For patient participants: usual care, as prescribed by the clinical care team, is unaffected by the study design and we only conduct observational measurements of patient participants during the course of the study.
  Interventions: Behavioral: Careverse

INTERVENTIONS:
Behavioral: Careverse — Careverse is a digital psychoeducational website designed to assist caregivers and patients to clarify their values, end-of-life preferences, enable surrogates to further their understanding of the patient's wishes, and prepare surrogates for the role and responsibilities of a medical decision maker. The intervention consists of values elicitation tools, educational materials, and testimonies. The participants will receive guides on how to initiate/re-introduce discussions about end-of-life wishes with their loved ones and clinicians.
  Arms: Intervention arm
Other: Usual Care — Caregivers in the comparator arm will receive a digital version of standard advanced care planning education material prepared by Agency of Integrated Care. The ACP Workbook is created by AIC to help individuals explore their values, care preferences, and end-of-life goals in a structured, reflective way.
  Arms: Comparator arm

SUMMARY:
The goal of this two-armed, parallel-design, pre-/post-intervention assessment clinical trial is to learn if a digital and interactive website helps to improve advance care planning (ACP) engagement among caregivers of patients with serious illness. The main questions it aims to answer are:

Does the website increase ACP engagement of caregivers of patients with serious illness? Researchers will compare the digital and interactive website to the usual care (a digital booklet) to see if the digital intervention works to improve ACP engagement among caregivers.

Participants who are caregivers will:

* Be introduced to a digital website and asked to explore the site over the course of the study.
* Complete four self-administered questionnaires (baseline, one-week, six-week, and six-month).

Participants who are patients will not have any intervention assigned and will only have their observational data collected through four interviewer-administered questionnaires (baseline, one-week, six-week, and six-month)

ELIGIBILITY:
1. Patient Participants Inclusion Criteria:

1. Singapore resident aged 21years and above,
2. patient able to identify one main caregiver in the care and medical decision-making for the patient;
3. patient able to communicate in either English, Chinese, Malay or Tamil;
4. patient meeting one of the following illness criteria: 4a. Patients with brain tumours: histological and/or radiological diagnosis of glioma or brain metastases.

4b. Patients with spontaneous intracerebral haemorrhage (SICH) based on radiological diagnosis of SICH on baseline computed-tomographic scans.

4c. Patients with CKD Stage 4 and 5, identified at G4 or G5 of CKD, glomerular filtration rate (GFR) 30 ml/min or less, inclusive of kidney failure on kidney replacement therapy; and (5) Physicians assessment that ACP is appropriate for the patient by physicians.* (*) The attending clinicians may base the assessment of ACP appropriateness on several factors in addition to high mortality risk. As a baseline, clinicians are asked to base their assessment of high mortality risk using the validated "Surprise" question.

2. Patient participants Exclusion Criteria:

1. Patients unable to identify a caregiver who is a medical decision-maker,
2. Patients are currently or was previously healthcare workers; or
3. Patients are diagnosed with dementia or deemed cognitively impaired as determined by the Abbreviated Mental Test.

3. Caregiver Participants Inclusion Criteria:

1. caregivers are identified as a medical decision-maker for the patient
2. Singapore resident aged 21 years and above; and
3. able to communicate in English

4. Caregiver Participants Exclusion Criteria:

1. caregivers are currently or were previously healthcare workers;
2. caregivers not involved in primary care of the patient (including providing care to the patient, supervision of care, or involved in making decisions regarding treatment the patient receives); or
3. caregivers diagnosed with dementia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Advance Care Planning Engagement Survey for Surrogate Decision-Maker | Baseline, 1-week, and 6-week
  The 17-item ACP Surrogate Decision Making Instrument (ACP-17 SDM) developed by Sudore et. al., is a validated questionnaire designed to assess how engaged surrogate decision makers (SDMs) are in the advance care planning process. The ACP-17 SDM measures engagement across three domains: 1) Serving as SDM (7 items), 2) Contemplation (4 items), and 3) Readiness (6 items). Each item is answered on a 5-point Likert scale (1 = not at all/never, to 5 = extremely/A lot), and higher mean scores (range: 1.0 - 5.0) indicate higher engagement in ACP by the surrogate.
  Van Scoy, Lauren J., et al. "Adaptation and preliminary validation of the advance care planning engagement survey for surrogate decision makers." Journal of pain and symptom management 57.5 (2019): 980-988.

SECONDARY OUTCOMES:
Satisfaction with care | Baseline, 6-week, and 6-month
  We measure patients and caregivers' satisfaction with care that they (or their patient) received using the Short Assessment of Patient Satisfaction (SAPS), a brief, validated, and generic 7-item questionnaire designed to efficiently measure patient satisfaction across a range of health care settings.[49-51] Each question is rated on a 5-point Likert scale (ranging from 0 to 4), and the items cover key domains of patient satisfaction including:1) Satisfaction with treatment, 2) Explanation of treatment results, 3) Clinician care and thoroughness, 4) Involvement in decision-making, 5) Respect received from the clinician, 6) Adequacy of time with the clinician, and 7) Overall satisfaction with care received. Total scores range from 0 to 28, and higher scores indicate greater satisfaction.
Satisfaction with care - Feeling Heard and Understood | Baseline, 6-week, and 6-month
  We measure how well patients and caregivers feel heard and understood by those caring for them in the hospital environment using the following point-of-care item: "Over the past 1(6) months, how much have you felt heard and understood by the doctors, nurses and hospital staff?". Response is rated on a 5-point scale (completely, quite a bit, moderately, slightly, not at all). Responses are reverse-coded, ranging from 1 - 5, with higher score indicates better quality of care.
  Gramling, R., et al., Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. Journal of Pain and Symptom Management, 2016. 51(2): p. 150-154.
Goals of care | Baseline, 1-week, 6-week, and 6-month
  We assess participants' preferences for aggressive care using goals of care questions adapted from the CanCORS Study. Participants were asked to trade-off between life-extension treatments or 1) those that miminise pain/discomfort and 2) those that were less costly. Participants responded on a scale of 1 to 9, where 1 represented maximal life extension with severe pain or discomfort (or with higher costs), 5 represented moderate life extension and moderate pain or discomfort (or moderate cost), and 9 indicated no life extension but minimal pain or discomfort (or lower costs). Scores 1 to 4 were categorized as prioritizing life extension, and scores 6 to 9 were categorized as prioritizing symptom management or cost containment.
  Malin, J.L., et al., Understanding cancer patients' experience and outcomes: development and pilot study of the Cancer Care Outcomes Research and Surveillance patient survey. Support Care Cancer, 2006. 14(8): p. 837-48.
Caregivers Wellbeing | Baseline, 1-week, 6-week, and 6-month
  We assess caregiver's quality of life using the Singapore Caregivers Quality of Life Scale (SCQOLS), a validated instrument developed specifically to assess the quality of life (QoL) of family caregivers of patients with advanced illnesses in Singapore. The 10-item SCQOLs measures five domains of quality of life of family caregivers of patients: (1) Physical Well-being (2 items); (2) Mental Well-being (2 items); (3) Experience & Meaning (2 items); (4) Impact on Daily Life (2 items) (5) Financial Well-being (2 items). Each item is rated on a 5-point scale, ranging from 0 (Not at All) to 4 (Very Much). Item scores are rescaled and summed. Total scores range from 0 - 100, with higher scores indicating better quality of life.
  Cheung, Yin Bun, et al. "Two valid and reliable short forms of the Singapore caregiver quality of life scale were developed: SCQOLS-10 and SCQOLS-15." Journal of Clinical Epidemiology 121 (2020): 101-108.
Caregiver quality of life - Mental health | Baseline, 1-week, 6-week, and 6-month
  Symptoms of depression and anxiety are measured using the 4-item Patient Health Questionnaire (PHQ-4), an ultra-brief, validated self-report instrument designed to screen for symptoms of both depression and anxiety in clinical and non-clinical populations. The PHQ-4 has four items: two for depression ("little interest or pleasure in doing things"; "feeling down, depressed, or hopeless") and two for anxiety ("feeling nervous, anxious or on edge"; "not being able to stop or control worrying"). Each item is rated based on symptom frequency over the past two weeks using a 4-point Likert scale, from 0 (not at all) to 3 (nearly every day). A subscale score of 3 or greater suggests possible anxiety or depression, while total distress is categorized as: normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Kroenke, K., et al., An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics, 2009. 50(6): p. 613-21.
Caregiver dyadic relationship | Baseline, 1-week, 6-week, and 6-month
  We assess the caregiving relationship between the caregiver and patient using the Dyadic Relationship Scale (DRS), a validated instrument measuring negative dyadic strain and positive dyadic interaction. [63] The caregiver version includes 11 items and are rated on a four-point scale (0 = strongly disagree to 3 = strongly agree). Total scores range from 0-33, with higher scores indicate better dyadic relationship.
  Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID: 18192628.
Patient Healthcare Utilisation | Within six months pre-and post-intervention OR 12 months before death
  Electronic medical records will be reviewed to find the number of inpatient admissions, urgent care visits, ED visits, hospitalizations, outpatient visits and aggressive treatment utilisation (e.g. Intubation, CPR, Surgery).
Patient quality of life | Baseline, 1-week, 6-week, and 6-month
  We assess patient's quality of life using the EQ-5D-5L instrument, a simple, and standardised measure of health status. five dimensions (mobility, self-care, usual activities, pain / discomfort and anxiety / depression), on five response levels: 1-no problems, 2-slight problems, 3-moderate problems, 4-severe problems, 5-unable to/extreme problems. The overall health states can be converted to an index value, ranging from 0 (worst possible health state) to 1 ((best possible health state) using a value set.
  Herdman, Michael, et al. "Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L)." Quality of life research 20.10 (2011): 1727-1736.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Choon Huat Koh, PhD(FM), Principal Investigator — Saw Swee Hock School of Public Health, National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The study gathers sensitive medical and personal data from patients and caregivers that cannot be disclosed publicly.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT07134881/Prot_SAP_000.pdf